CLINICAL TRIAL: NCT03998826
Title: Effect of Piroxicam Premedication on Postendodontic Pain in Mandibular Molars With Non-vital Pulp: A Randomized Controlled Trial
Brief Title: Piroxicam Premedication for Postendodontic Pain in Non-vital Mandibular Molars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Asmaa Fathelrahman Mohamed, Postgraduate Student, Department of Endodontics, Faculty of Dentistry, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CEBD-CU-2019-06-13
Record Dates: First submitted 2019-06-25; First posted 2019-06-26 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Non-Vital Tooth
Keywords: Piroxicam; Postendodontic pain; analgesic intake
MeSH Terms: conditions — Tooth, Nonvital | interventions — Piroxicam

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Type: Two arm, parallel, randomized clinical trial. Allocation ratio: 1:1 Framework: Superiority.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study will be participant and operator-blind where the participant and operator will not know the intervention done.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Piroxicam drug (Experimental): 20 mg piroxicam
  Interventions: Drug: Piroxicam
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Piroxicam — 20mg piroxicam
  Arms: Piroxicam drug
Drug: Placebo — placebo
  Arms: Placebo

SUMMARY:
The aim of the study is to evaluate the effect of piroxicam (20mg) compared to placebo on post-endodontic pain of single-visit endodontic treatment of non-vital mandibular molars.

DETAILED DESCRIPTION:
* Patients will be clinically and radiographically examined and their eligibility will be assessed. Eligible patients will be treated in one visit.
* Patients will be randomly assigned to one of 2 groups: experimental group (premedication with 20 mg of piroxicam) and the control group (premedication with placebo). Each participant will receive a standard inferior alveolar nerve block injection. After endodontic treatment, patients will be given postoperative instructions and informed, in case of pain, to receive ibuprofen 200 mg as rescue medication.
* Postendodontic pain intensity and incidence at the different pain categories (No, mild, moderate, severe) will be assessed 6, 12, 24, 48, 72 hours and 7 days postoperatively using a 0-10 numerical rate scale (NRS). Analgesic intake throughout the 7 days will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aging between 18-50 years old
2. Patients with mandibular molar with non-vital pulp.
3. Systemically- healthy patients (ASA I or II).
4. Patients who agree to attend for recall appointments and provide a written consent.

Exclusion Criteria:

1. Pregnant or lactating female patients.
2. Patients allergic to piroxicam.
3. History of peptic ulceration.
4. Periapical abscess, fistula.
5. Non-restorable teeth.
6. Moderate or severe marginal periodontitis i.e. pocket probe>3mm.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Postendodontic pain using a pain-measuring scale | 6 hours
  Postoperative pain is measured using the Numerical Rating Scale (NRS) which is an 11-point scale from 0-10 where 0 represents no pain and 10 represents the worst pain measured 6 hours after the first visit
Postendodontic pain using a pain-measuring scale | 12 hours
  Postoperative pain is measured using the Numerical Rating Scale (NRS) which is an 11-point scale from 0-10 where 0 represents no pain and 10 represents the worst pain measured 12 hours after the first visit
Postendodontic pain using a pain-measuring scale | 24 hours
  Postoperative pain is measured using the Numerical Rating Scale (NRS) which is an 11-point scale from 0-10 where 0 represents no pain and 10 represents the worst pain measured 24 hours after the first visit
Postendodontic pain using a pain-measuring scale | 48 hours
  Postoperative pain is measured using the Numerical Rating Scale (NRS) which is an 11-point scale from 0-10 where 0 represents no pain and 10 represents the worst pain measured 48 hours after the first visit
Postendodontic pain using a pain-measuring scale | 72 hours
  Postoperative pain is measured using the Numerical Rating Scale (NRS) which is an 11-point scale from 0-10 where 0 represents no pain and 10 represents the worst pain measured 72 hours after the first visit
Postendodontic pain using a pain-measuring scale | 7 days
  Postoperative pain is measured using the Numerical Rating Scale (NRS) which is an 11-point scale from 0-10 where 0 represents no pain and 10 represents the worst pain measured 7 days after the first visit

SECONDARY OUTCOMES:
Analgesic medication intake incidence | 7 days
  Analgesic medication intake incidence (Yes/No) as a rescue medication in case postoperative pain persisted after the sham medication intake.

CONTACTS AND LOCATIONS:
Overall Officials: Asmaa FE Mohamed, B.D.S, Principal Investigator — Cairo University

REFERENCES:
- [Background] Konagala RK, Mandava J, Pabbati RK, Anupreeta A, Borugadda R, Ravi R. Effect of pretreatment medication on postendodontic pain: A double-blind, placebo-controlled study. J Conserv Dent. 2019 Jan-Feb;22(1):54-58. doi: 10.4103/JCD.JCD_135_18. PMID 30820083
- [Background] Joshi N, Mathew S, George JV, Hegde S, Bhandi S, Madhu KS. Comparative evaluation of the efficacy of two modes of delivery of Piroxicam (Dolonex((R))) for the management of postendodontic pain: A randomized control trial. J Conserv Dent. 2016 Jul-Aug;19(4):301-5. doi: 10.4103/0972-0707.186454. PMID 27563175
- [Background] Nekoofar MH, Sadeghipanah M, Dehpour AR. Evaluation of meloxicam (A cox-2 inhibitor) for management of postoperative endodontic pain: a double-blind placebo-controlled study. J Endod. 2003 Oct;29(10):634-7. doi: 10.1097/00004770-200310000-00005. PMID 14606784
- [Derived] Mohamed AF, El-Asfouri HA, Amin SAW. Effect of sublingual fast-dissolving piroxicam premedication on postoperative pain experience in mandibular molars with non-vital pulp: a randomized double-blind controlled trial. Head Face Med. 2024 Sep 21;20(1):52. doi: 10.1186/s13005-024-00453-x. PMID 39306665